CLINICAL TRIAL: NCT04082468
Title: Observational Trial Evaluating Whether Elevated Factor VIII Activity During Multiple Sclerosis Relapses Serves as a Marker for Solumedrol-Resistance and Incomplete Relapse Recovery
Brief Title: VALIDATE: Factor VIII Trending for MS Relapse
Status: Withdrawn | Type: Observational
Why Stopped: Never started enrollment due to logistics.
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Responsible Party: Sponsor
Other Study IDs: 18-500-440-30-10
Record Dates: First submitted 2019-09-05; First posted 2019-09-09 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Multiple Sclerosis
Keywords: Relapsing remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting | interventions — Bleeding Time

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Blood sample collection for coagulation profile — Factor VIII Activity Level, Factor VIII Antigen Level, Interleukin 6, vWF Antigen Level, Thrombin Activity, Protein C Activity, Protein C Antigen Level, CRP, PT/PTT/INR ,T & B lymphocyte panel at above time points
  Other Names: Clinical data collection

SUMMARY:
Multiple sclerosis (MS) patients hospitalized with an acute motor or visual relapse will be consented. Factor VIII-related labs will be systematically drawn for six months. During this time, patients will be followed with clinical assessments including: Expanded Disability Status Scale (EDSS), Multiple Sclerosis Functional Composite (MSFC), Low Contrast Sloan Letter Chart Testing, Symbol Digital Modality Test (SDMT), and NeuroQol. MRIs of the brain, cervical spine, and thoracic spine with and without contrast will be obtained. All patients will be treated with 1 gram IV solumedrol daily for five days per standard care. Clinical, imaging, and Factor VIII-related lab data individually or in aggregate will be correlated with relapse presence, severity, and extent of recovery following standard intravenous (IV) solumedrol treatment

DETAILED DESCRIPTION:
The identification of blood tests that detect patients having Multiple Sclerosis (MS) relapses in real time could lead to a new era of MS relapse treatment. Accidental, anecdotal clinical observations suggest that transient upregulation of the intrinsic coagulation pathway, namely with elevated von Willebrand Factor antigen levels (vWF) and increased Factor VIII activity, occur with some MS relapses and that the higher the elevated plasma values, the more glucocorticoid therapy required to achieve clinical improvement.

Ten adult patients with relapsing remitting MS with or without secondary progression will be consented and enrolled in this longitudinal clinical trial. As a standard of care all patients will be treated daily with one gram IV solumedrol for five days, and all patients will have performed standard MRI's of the brain, cervical spine, and thoracic spine with and without IV contrast during hospital admission, which may occur after Solumedrol treatment.

In addition to this standard of care, patients will have a panel of labs drawn on Days: 1 (prior to any solumedrol treatment), 7, 15, 30, 45, 60, 90, 135, and 180. Neurological clinical assessments, comprising of assessing the EDSS score, the MSFC index (that looks at ambulation, hand/arm coordination, and cognitive function, comprised of the 25 foot timed walking tests, with and without any assistive devices if possible), LCSLC test, SDMT, and Neuro QoL will be conducted on Days: 1, 7, 30, 90, 180. Individual and aggregate laboratory values, neurological clinical assessment results, and MRI findings will be correlated for the presence of a MS relapse, severity of relapse, and extent of recovery from the relapse. Patients and evaluators will be blinded to the lab results.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged 18-65 with an established diagnosis of relapsing remitting multiple sclerosis (RRMS);
2. Patients with RRMS hospitalized at St. Joseph's Hospital and Medical Center in Phoenix, Arizona for an acute relapse affecting strength or vision;
3. Patients may or may not be on disease modifying treatment;
4. Entry EDSS score up to 7.0.

Exclusion Criteria:

1. Patients unable to have an MRI;
2. Patients taking any heparin products, warfarin (Coumadin), apixiban (Eliquis), dabigatran (Pradaxa), or rivaroxaban (Xarelto);
3. If stroke, tumor or other non-MS related cause is identified as the source of the patient's neurological issues.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute MS relapse patients hospitalized at St. Joseph's Hospital and Medical Center in Phoenix, Arizona
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-08-13 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Correlation of MS relapse recovery time with elevated lab values. | 180 days
  Extent of relapse recovery across a variety of measures will be correlated with collected lab values and neurological assessments in an attempt to identify a positive correlation between incomplete recovery and solumedrol resistance with abnormally elevated lab values involving the vWF antigen and Factor VIII pathways

CONTACTS AND LOCATIONS:
Overall Officials: Amiee Borazanci, MD, Principal Investigator — St. Joseph's Hospital/Barrow Neurological Institute
Locations (1):
- Barrow Neurological Institute, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No